CLINICAL TRIAL: NCT03595813
Title: Identifying Immune-related Biomarkers to Predict the Efficacy of Cancer Immunotherapy-IMMUNO-SUP-IPC 2017-002
Brief Title: Identifying Immune-related Biomarkers to Predict the Efficacy of Cancer Immunotherapy
Acronym: IMMUNO-SUP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Cancer Research Center of Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IMMUNO-SUP-IPC 2017-002
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer Metastatic; Locally Advanced Malignant Neoplasm; Non Hodgkin Lymphoma; Urologic Neoplasms
Keywords: Immune check point blockade; biomarkers; immunomonitoring
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Urologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with Immune Checkpoint Blockade (Experimental)
  Interventions: Procedure: Blood sample collection; Procedure: Biopsy collection

INTERVENTIONS:
Procedure: Blood sample collection — Blood samples collection (5EDTA vials) at baseline, post infusion of ICB n°2/4/8 and at progression
Procedure: Biopsy collection — Optional biopsy collection at baseline and progression

SUMMARY:
The development of Immune Checkpoint Blockade (ICB) is a revolution in medical oncology as ICB have changed the standard treatments of several metastatic tumor types. However, the response rate to ICB is low, and the biological bases for this response heterogeneity are poorly understood.

In the frame of Immunosup study, we will collect blood (at baseline, post infusion of ICB n°2/4/8 and at progression) and tumor samples (optional: at baseline and progression) from patients with locally advanced or metastatic cancer, treated with ICB, in order to determine if the dynamics of immunosuppressive actors (MDSC, TReg, Immunosuppressive cytokines) predicts response to these immunotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of locally advanced or metastatic solid tumor or lymphoma treated with Immune check blockade
* Signed informed consent
* Affiliated to(or beneficiary of) the French Social Security

Exclusion Criteria:

* Pregnant or breastfeeding woman or woman who does not apply effective contraception
* Emergency
* Vulnerable person or unable to provide informed consent
* Emergency
* Person unable to comply with required study follow up
* Contraindication to the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Plasma immunosuppressive actors in patients treated with a Checkpoint inhibitor | 4 months
  Measure (by flux cytometry) and comparison of plasma immunosuppressive actors, between baseline and the 4th injection of an Immune Checkpoint inhibitor

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli-Calmettes, Marseille, Bouches-du-Rhône, France